CLINICAL TRIAL: NCT07106554
Title: Impact of Holotropic Breathwork on Nursing Student Mental Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment lower than expected
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0034-24-FB
Record Dates: First submitted 2025-07-18; First posted 2025-08-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Mental Health
Keywords: holotropic breathwork; nursing student; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- holotropic breathwork (Experimental): participants will experience holotropic breathwork
  Interventions: Behavioral: holotropic breathwork

INTERVENTIONS:
Behavioral: holotropic breathwork — participants will engage in holotropic breathwork

SUMMARY:
Purpose of the Study

This study investigates whether Holotropic Breathwork (HB)-a technique involving controlled hyperventilation paired with music and guided support-can improve the mental, emotional, and existential well-being of nursing students. The researchers aim to:

Evaluate the acceptability and impact of HB in this population.

Compare psychological, interpersonal, and existential functioning before and after the breathwork session.

Study Design Participants: Up to 72 current UNMC nursing students (age 19+), excluding those with bipolar/psychotic disorders, cardiac/seizure conditions, glaucoma, or recent surgeries. Pregnant individuals are excluded.

Intervention: A single-day breathwork session, led by certified facilitators, including preparatory instruction, two breathwork rounds (one as "breather," one as "sitter"), and integration discussions.

Data Collection: Surveys before, immediately after, and at 1-, 3-, and 6-month follow-ups. Instruments include:

Patient Health Questionnaire-9 (PHQ-9)

General Anxiety Disorder-7 (GAD-7)

Psychological Insight Scale

Self and Interpersonal Functioning Scale

Purpose in Life Test

Emotional Breakthrough and Mystical Experience Questionnaires

Significance Nursing students face significant stress, anxiety, and even suicide risk. HB may offer a safe, non-drug intervention to support their mental health. While HB has been studied in other populations, this is the first known study targeting nursing students.

Safety Measures Participants monitored by trained facilitators.

Pre-screening includes a urine pregnancy test.

Emergency plans include psychiatric assessment, Uber/Lyft rides if needed, and referral systems for mental health support.

If >15% of participants experience serious adverse events, the study will be halted.

DETAILED DESCRIPTION:
Study design overview The study is a non randomized interventional pilot trial assessing whether a single day of Holotropic Breathwork (HB) improves mental health among University of Nebraska Medical Center (UNMC) nursing students. Holotropic Breathwork involves self directed hyperventilation while lying down, accompanied by music and trained facilitators. HB has been studied among the general public and patients with substance use disorders, but it has not been trialed among nursing students. The study will examine changes in mystical experiences, challenging experiences, emotional breakthroughs and psychological insight (Aim 1) and will compare pre and post HB psychological, interpersonal and existential functioning (Aim 2). Up to 70 students will be enrolled (two sessions with ≤30 participants each). All sessions will take place at the UNMC College of Nursing in Lincoln.

Intervention

Participants will attend a day long HB workshop. Each workshop is led by at least two certified facilitators and two apprentices. The workshop follows a structured sequence:

* Opening circle and orientation: Participants introduce themselves and share their motivation. Facilitators give a 60 minute presentation covering the concept of the inner healer, the difference between holotropic and hylotropic states, a historical overview of altered states of consciousness, how HB was developed, and practical tips for the session. Participants agree to confidentiality, to remain on site until dismissed, and to avoid harming themselves or others. Facilitators explain the roles of "sitter" and "breather".
* Partner assignment: Each student chooses a partner. If pairs cannot be formed, facilitators assist; groups with two breathers and one sitter can be accommodated.
* Breathwork session (first group): The breather lies on a mat wearing eye shades. After a guided relaxation, participants gradually begin deep, rapid breathing. They may adjust the pace as needed. Purposefully selected music plays for two to three hours. Responses vary: some lie still, others move or vocalize. Sitters provide support (tissues, water, walking to the restroom) and avoid interfering unless requested. Facilitators manage the music, ensure safety and intervene only at the participant's request. At least two facilitators and apprentices maintain a 1 : 5 breather to staff ratio.
* Break and lunch: After the first breathwork session, facilitators conduct short one on one check ins to ensure participants feel ready to rejoin the group. A light lunch is served.
* Second breathwork session with role reversal: Partners switch roles so that the previous sitter experiences breathwork.
* Integration presentation: After both sessions, facilitators deliver a second 60 minute presentation on integration and self care. They explain formal and informal integration, self care practices, and recommend delaying major life decisions until after participants have time to reflect.
* Closing circle: Participants share their experiences without receiving feedback. Those needing additional processing can meet privately with a facilitator. Before leaving the campus, participants complete the post experience survey.

Participant eligibility

* Inclusion criteria: Current UNMC nursing students (bachelor's, master's or doctoral level) ≥19 years old.
* Exclusion criteria: Students will be excluded if they self report any of the following: bipolar disorder or psychotic disorder; lifetime psychotic symptoms; cardiac conditions or current cardiac symptoms; history of seizure disorder; uncontrolled hypertension ≥140/90 mm Hg; glaucoma or retinal detachment; recent surgeries; pregnancy. The study specifically excludes pregnant women and verifies absence of pregnancy with a CLIA waived urine test on the morning of breathwork. Women of child bearing potential are included without contraception requirements because pregnancy status is verified immediately before the intervention.

Recruitment procedures Recruitment begins with the principal investigator (PI) sending an email to UNMC nursing students describing the opportunity to participate. Interested students contact the PI via email. A follow up email contains links to two YouTube videos explaining Holotropic Breathwork; students are asked to watch the videos and then email the PI again if they remain interested. The PI schedules an informed consent meeting in person or via Zoom. During this meeting, the PI describes the HB process, answers questions, confirms understanding and obtains consent in person or via DocuSign.

Approximately one week before the breathwork day, participants receive a REDCap baseline survey that collects demographic data (sex, age, program of study) along with the Patient Health Questionnaire 9 (PHQ 9), Generalized Anxiety Disorder 7 (GAD 7), Self and Interpersonal Functioning Scale (SIFS) and Purpose in Life Test - Short Form (PIL SF). Students with asthma are instructed to bring an inhaler; those experiencing an asthma attack during breathwork may continue if the inhaler resolves symptoms.

Data collection schedule

Data are collected at multiple time points:

Timing / Assessment Measures Purpose Baseline (≈1 week prior) Demographics, PHQ 9, GAD 7, SIFS, PIL SF Characterize participants and pre intervention mental health Day of breathwork (morning) Urine pregnancy test (for those of child bearing potential); blood pressure screening for uncontrolled hypertension Safety screening Immediately after breathwork Mystical Experiences Questionnaire, Challenging Experiences Questionnaire, Emotional Breakthrough Inventory and Psychological Insight Scale Evaluate acute subjective experiences

1, 3 and 6 months post HB Psychological Insight Scale, PHQ 9, GAD 7, SIFS and PIL SF Measure sustained changes in psychological, interpersonal and existential functioning Safety and risk monitoring The PI reviews each completed PHQ 9 within one hour (8 AM - 10 PM) or by 9 AM the next morning and takes appropriate action. If a score >14 and suicidal ideation (question 9) are reported, the PI contacts the participant by phone and email and arranges for emergency evaluation; if no response is received within 30 minutes, local authorities perform a welfare check. High PHQ 9 scores without suicidal ideation prompt a mental health consultation; suicidal ideation with lower scores prompts assessment and referral. Participants who are unsteady at the end of the day receive a ride home via Lyft or Uber and, if needed, a return ride the next day. Participants experiencing a medical event during breathwork are withdrawn from the study. To reduce risk, all participants agree not to harm themselves or others and to remain on site until released. The presence of certified facilitators and apprentices ensures a supportive ratio (~1 : 5) and that no breather is left alone. Students with asthma must bring an inhaler; if an asthma attack occurs and is resolved, the participant may continue.

Integration and follow up Immediately after both breathwork sessions, facilitators deliver an integration presentation covering formal and informal methods, self care practices (e.g., relaxation, art, journaling) and strategies for processing the experience before making major decisions. A closing circle allows participants to share reflections without feedback. Those needing further processing can meet privately with a facilitator. Unlike the group activities protocol for individuals with substance use disorders, there are no additional Zoom based integration groups; follow up focuses solely on completing REDCap surveys at 1, 3 and 6 months.

Participant location and resources All sessions and consent meetings take place at the UNMC College of Nursing in Lincoln, Nebraska. The college provides large rooms suitable for both informed consent meetings and breathwork exercises. Data are stored securely in UNMC's Microsoft 365 environment and REDCap database. Confidential identifiers such as names and email addresses are recorded to link survey data. Statistical analysis will use paired samples t tests to compare pre and post HB survey results, with more complex models applied as the data allow.

Summary This protocol outlines a structured, single day holotropic breathwork intervention for nursing students. By combining careful screening, thorough orientation, a controlled breathing experience with professional facilitation, and multiple assessments over six months, the study aims to determine the acceptability and impact of HB on students' psychological, interpersonal and existential functioning. Safety is addressed through rigorous exclusion criteria, pregnancy and blood pressure screening, monitoring of mental health scores and provision of transportation when necessary. The results will inform whether HB could serve as a novel, adjunctive approach to support nursing student mental health.

ELIGIBILITY:
Inclusion Criteria:

- Currently enrolled in a program at the UNMC College of Nursing (bachelor's, master's, or doctorate).

19 years of age or older.

Exclusion Criteria:

* Diagnosed with bipolar disorder at any point in life (per self-report).

Diagnosed with a psychotic disorder or have experienced psychotic symptoms at any point in life (per self-report).

Diagnosed with a cardiac condition, received care for a cardiac condition, or currently have cardiac symptoms (per self-report).

Ever diagnosed with a seizure disorder (per self-report).

Uncontrolled hypertension, defined as 140/90 mmHg or greater (measured the morning of the breathwork).

Diagnosed with glaucoma or retinal detachment.

Recent surgeries (unspecified, but likely judged as too recent for safe participation).

Currently pregnant (verified with a urine pregnancy test the morning of the breathwork).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | 6 months
  PHQ-9, 0 - 27 Higher scores indicate more severe depressive symptoms. Scores classify depression severity (e.g., 0 4 no/minimal, 20 27 severe).
Generalized Anxiety Disorder-7 | 6 months
  0 - 21 Higher scores represent more severe anxiety. Scores of 0 4 = minimal, 5 9 = mild, 10 14 = moderate and 15 21 = severe.
Psychological Insight Scale | 6 months
  6 - 42 (6 items × 1-7) Higher scores denote greater psychological insight and a higher likelihood of meaningful psychological or behavioral change.
Self and Interpersonal Functioning Scale | 6 months
  0 - 96 (24 items × 0-4) Higher scores indicate greater dysfunction (worse personality/self interpersonal functioning).
Purpose in Life Test | 6 months
  6 - 42 (6 items × 1-7) After reverse scoring, higher summed scores represent greater psychological well being and a stronger sense of purpose.
Emotional Breakthrough Inventory | 6 months
  0 - 600 (6 items × 0-100) Higher scores indicate a greater emotional breakthrough, reflecting the extent of emotional release or resolution.
Mystical Experience Questionnaire | 6 months
  0 - 150 (30 items × 0-5) Higher scores indicate a more intense mystical or spiritual experience.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Medical Center, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No